CLINICAL TRIAL: NCT01668953
Title: Impact of Platelet Rich Plasma Over Alternative Therapies in Patients With Lateral Epicondylitis
Brief Title: Comparison of Platelet Rich Plasma and Alternative Therapies for the Treatment of Tennis Elbow (Lateral Epicondylitis)
Acronym: IMPROVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not analyze data
Sponsor: McMaster University (Other)
Collaborators: Arthrex, Inc. (Industry); The Physicians' Services Incorporated Foundation (Other); Radiological Society of North America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMPROVE-001; Research Seed Grant # 1204 (Other Grant/Funding Number: Radiological Society of North America (RSNA)); NCT01789632 (obsolete NCT alias)
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Lateral Epicondylitis (Tennis Elbow)
Keywords: Lateral Epicondylitis; Tennis Elbow; Platelet Rich Plasma; Whole Blood; Tendon Fenestration
MeSH Terms: conditions — Tennis Elbow | interventions — Injections; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Platelet Rich Plasma (PRP) Injection (Experimental): Patients in this arm will receive a platelet rich plasma injection at the site of their lateral epicondylitis, followed by post-treatment physical therapy exercises.
  Interventions: Other: Platelet Rich Plasma (PRP) Injection
- Whole Blood Injection (Active Comparator): Patients in this arm will receive a whole blood injection at the site of their lateral epicondylitis, followed by post-treatment physical therapy exercises.
  Interventions: Other: Whole Blood Injection
- Dry Needle Fenestration (Active Comparator): Patients in this arm will receive 15-25 gentle strokes of dry needling (piercing of the tendon) at the site of their lateral epicondylitis, followed by post-treatment physical therapy exercises. No blood will be injected into the tendon.
  Interventions: Other: Dry Needle Fenestration
- Sham Injection (Placebo Comparator): Patients in this arm will receive a sham injection, followed by post-treatment physical therapy exercises. No blood will be injected into the tendon.
  Interventions: Other: Sham Injection

INTERVENTIONS:
Other: Platelet Rich Plasma (PRP) Injection — 1. The subcutaneous soft tissues of the lateral elbow will be infiltrated with 1% lidocaine for local anesthetic.
  2. A 22-gauge needle will then be placed into the tendon followed by 15-25 gentle strokes of dry needling in which the needle pierces the tendon at multiple sites.
  3. For the PRP preparation, the Arthrex ACP system will be used. This is a closed, double syringe system which uses 16 mL of whole blood drawn from the patient's contralateral arm, using a 19G butterfly needle. The blood is centrifuged at 1500 rpm for 5 minutes and extracts 4-7 ml of PRP. No anticoagulant will be used.
  4. Fenestration of the tendon will continue as 3mL of PRP is injected into the common extensor tendon.
  5. The remaining PRP will be sent for analysis of platelet, WBC, and RBC concentrations.
  Arms: Platelet Rich Plasma (PRP) Injection
Other: Whole Blood Injection — 1. The subcutaneous soft tissues of the lateral elbow will be infiltrated with 1% lidocaine for local anesthetic.
  2. A 22-gauge needle will then be placed into the tendon followed by 15-25 gentle strokes of dry needling in which the needle pierces the tendon at multiple sites.
  3. 6mL of autologous whole blood will be drawn from the patient's contralateral arm, using a 19G butterfly needle.
  4. Fenestration of the tendon will continue as 3mL of whole blood biologic agent is injected into the common extensor tendon.
  5. The remaining 3mL will be sent for analysis of platelet, WBC, and RBC concentrations.
  Arms: Whole Blood Injection
Other: Dry Needle Fenestration — 1. The subcutaneous soft tissues of the lateral elbow will be infiltrated with 1% lidocaine for local anesthetic.
  2. 3mL of autologous whole blood will be drawn from the patient's contralateral arm, using a 19G butterfly needle, and discarded.
  3. A 22-gauge needle will then be placed into the tendon.
  4. 15-25 strokes or as many strokes required until tendon is softened of dry needling will be performed in which the needle pierces the tendon at multiple sites. No blood will be injected into the tendon.
  Arms: Dry Needle Fenestration
Other: Sham Injection — 1. The subcutaneous soft tissues of the lateral elbow will be infiltrated with 1% lidocaine (no epinephrine) for local anesthetic.
  2. 3mL of autologous whole blood will be drawn from the patient's contralateral arm, using a 19G butterfly needle, and discarded.
  3. The superficial subcutaneous soft tissues will be re-entered however, the tendon itself will not be entered and nothing will be injected.
  Arms: Sham Injection

SUMMARY:
"Tennis elbow" is the most common cause of lateral elbow pain, generally caused by either work or sports related repetitive strain. In this condition, a tendon along the outside of the elbow becomes inflamed leading to pain, especially with flexing and extending the elbow.

Many treatments have been attempted, including physiotherapy and steroids, with little success. One treatment which has been very effective is the injection of the patients own blood (taken from their other non-affected arm) into their abnormal tendon. The blood recruits the patients own healing factors and heals the damaged tendon. As platelets are thought to be largely responsible, injection of concentrated platelets, extracted from the patient's blood (platelet rich plasma) is a newer, but expensive, technique.

At this point, it is unclear whether whole blood, concentrated platelets, or simply passing a ultrasound-guided needle through the abnormal tendon as a means to stimulate tissue healing (tendon fenestration) is the better treatment.

The objective of this trial is to compare platelet rich plasma, whole blood, dry needle tendon fenestration, and sham injection (with physical therapy) to identify the best and most cost-effective therapy for this debilitating condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult man or woman aged 18 years or greater.
* Clinical diagnosis of lateral epicondylitis based on site of pain, pain elicited with active extension of the wrist in pronation and elbow extension.
* Documented sonographic diagnosis of common extensor tendinosis based on tendon thickening, areas of hypoechogenicity, and loss of the normal echotexture.
* Chronic symptoms (equal or greater than 3 months).
* Pain of at least 5 out of 10 on a visual analog scale (VAS).
* Provision of informed consent.

Exclusion Criteria:

* Acute symptom onset (less than 2 months).
* History of acute elbow trauma (less than one week).
* History of rheumatoid arthritis.
* History of malignancy.
* Pregnancy
* Patients requiring anti-platelet medication for the treatment of heart attack, stroke or other medical condition.
* Previous surgery for lateral epicondylitis.
* Previous local injections, including steroids within the past 6 months.
* Signs of other causes for lateral elbow pain (posterior interosseous nerve entrapment, osteochondral lesion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-08; Primary Completion 2023-04 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
Pain Reduction | Baseline, 6 weeks, 3, 6, 12 months
  Pain reduction will be measured using the Visual Analog Scale (VAS), a subjective scale in which the patient rates their pain on a scale from 0 to 10 (0, no pain, 10, maximum possible pain).

SECONDARY OUTCOMES:
Functional Disability | Baseline, 6 weeks, 3, 6, 12, 24 months
  Functional disability will be measured using the Liverpool Elbow Score (LES) which is an assessment tool for evaluating function based on range of motion, ulnar nerve function, and ability to perform daily activities.
Psychological Impairment | Baseline, 6 weeks, 3, 6, 12, 24 months
  Psychological impairment (depression and anxiety) will be assessed using the Hospital Anxiety and Depression Scale (HADS) which is a reliable, validated, and practical tool for identifying and quantifying anxiety and depression.
Health-Related Quality of Life | Baseline, 6 weeks, 3, 6, 12, 24 months
  Health-related quality of life will be measured using the 12-Item Short Form Health Survey (SF-12).

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Chiavaras, MD, PhD, Principal Investigator — McMaster University
Locations (2):
- University of Michigan, Ann Arbor, Michigan, United States
- Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Karjalainen TV, Silagy M, O'Bryan E, Johnston RV, Cyril S, Buchbinder R. Autologous blood and platelet-rich plasma injection therapy for lateral elbow pain. Cochrane Database Syst Rev. 2021 Sep 30;9(9):CD010951. doi: 10.1002/14651858.CD010951.pub2. PMID 34590307